CLINICAL TRIAL: NCT05750745
Title: A 12-Week, Randomised, Controlled, Examiner-blind, Clinical Study to Evaluate the Efficacy of a Stannous Fluoride Toothpaste for the Relief of Dentine Hypersensitivity in a Chinese Population
Brief Title: A Clinical Study to Evaluate the Efficacy of a Stannous Fluoride Toothpaste for the Relief of Dentine Hypersensitivity in a Chinese Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 300026
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Results first posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-09

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Chewing Gum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test Dentifrice (Experimental): Participants will be instructed to brush the two test teeth first, then the whole mouth (all teeth) for 1-timed minute, twice daily (morning and evening) with Sensodyne Sensitivity & Gum. After brushing, participants will be instructed to rinse once with 10 milliliters (mL) of water using the measuring cup provided.
  Interventions: Drug: Sensodyne Sensitivity & Gum
- Negative Control (Active Comparator): Participants will be instructed to brush the whole mouth (all teeth) for 1-timed minute, twice daily (morning and evening) with Crest Cavity Protection Fresh Lime. After brushing, participants will be instructed to rinse once with 10 mL of water using the measuring cup provided.
  Interventions: Drug: Crest Cavity Protection Fresh Lime
- Positive Control (Active Comparator): Participants will be instructed to brush the whole mouth (all teeth) for 1-timed minute, twice daily (morning and evening) with Sensodyne Repair and Protect. After brushing, participants will be instructed to rinse once with 10 mL of water using the measuring cup provided.
  Interventions: Drug: Sensodyne Repair and Protect

INTERVENTIONS:
Drug: Sensodyne Sensitivity & Gum — Sensodyne Sensitivity & Gum toothpaste is containing 0.454% w/w SnF2.
  Arms: Test Dentifrice
Drug: Crest Cavity Protection Fresh Lime — Crest Cavity Protection Fresh Lime is containing 1150 parts per million (ppm) fluoride as Sodium fluoride (NaF).
  Arms: Negative Control
Drug: Sensodyne Repair and Protect — Sensodyne Repair and Protect toothpaste is containing 5.0% w/w calcium sodium phosphosilicate (CSPS).
  Arms: Positive Control

SUMMARY:
The purpose of this study is to evaluate the efficacy of the 0.454 percentage (%) weight/weight (w/w) stannous fluoride (SnF2) toothpastes for the relief of dentine hypersensitivity (DH) in China.

DETAILED DESCRIPTION:
This study will be a single center, randomized, controlled, examiner-blind, 3 treatment arm, parallel group design study, stratified by maximum baseline Schiff sensitivity score (of the 2 selected 'test teeth'), with a treatment period of 12 weeks, to investigate the clinical efficacy of a SnF2 toothpaste for the relief of DH in a Chinese population. The SnF2 test dentifrice will be compared to commercialized negative and positive control toothpastes.

ELIGIBILITY:
Inclusion Criteria:

* Participant provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any study procedures are performed.
* Participant who is willing and able to understand and comply with scheduled visits, product usage requirements and other study procedures.
* A participant in good general, oral and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant or relevant abnormalities in medical history or upon oral examination, or condition, that would impact the participant's safety, wellbeing or the outcome of the study, if they were to participate in the study, or affect the individual's ability to understand and follow study procedures and requirements.
* Participant who owns a smartphone with the WeChat application installed.
* A participant who presents the following oral and dental inclusions will apply at Screening (Visit 1):

  1. Self-reported history of tooth sensitivity lasting more than six months but not more than 10 years and experience DH symptoms at least 'once a week' or more frequently (as mentioned in Screening questionnaire).
  2. Good general oral health, with a minimum of 20 natural teeth.
  3. Minimum of 2 accessible non-adjacent teeth (incisors, canines, pre-molars), preferably in different quadrants, with clinically confirmed DH.
* Each eligible tooth must meet all of the following criteria:

  1. Exposed dentine due to facial/cervical erosion, abrasion or gingival recession (EAR).
  2. Modified Gingival Index (MGI) = 0 directly adjacent to the exposed dentine (i.e., the test area) only
  3. Clinical mobility = 0.
  4. DH as evidenced by qualifying levels of tactile and evaporative (air) sensitivity (tactile threshold less than or equal to [<=] 20 g and Schiff sensitivity score more than or equal to [>=] 2).
* A participant who presents the following oral and dental inclusions will apply at Baseline (Visit 2):
* All teeth identified at Screening (Visit 1) as eligible for Baseline assessments will be reassessed for tactile sensitivity first; eligible teeth with Baseline tactile threshold <= 20g will then be re-assessed for evaporative (air) sensitivity.
* Participants must have a minimum of two non-adjacent, accessible teeth (incisors, canines, pre-molars), preferably in different quadrants, with clinically confirmed DH as evidenced by qualifying levels of tactile and evaporative (air) sensitivity:

  1. Tactile threshold <= 20 g at Screening and Baseline
  2. Schiff sensitivity score >= 2 at Screening and Baseline.
  3. VAS >= 40 mm at Baseline.
* The clinical examiner will select two 'test teeth' from those eligible teeth which meet the tactile threshold and Schiff sensitivity score criteria at both Screening and Baseline, and the VAS criterion at Baseline.
* Each test tooth must demonstrate a consistent DH response to the evaporative (air) stimulus at both Screening and Baseline:

  1. Screening Schiff sensitivity score = 2 and Baseline Schiff sensitivity score = 2 or Screening Schiff sensitivity score = 3 and Baseline Schiff sensitivity score = 3.

Exclusion Criteria:

* Participant who is an employee of the study site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the study site otherwise supervised by the investigator; or a sponsor employee directly involved in the conduct of the study or a member of their immediate family.
* Participant who has participated in, or has participated in, other studies (including non-medicinal studies) involving investigational product(s) within 30 days of Screening (Visit 1).
* Participant who is participating in, has participated in, a study evaluating a tooth desensitizing treatment within 8 weeks of Screening (Visit 1).
* Participant who is using, or has used, an oral care product indicated for DH relief within 8 weeks of Screening (Visit 1). Participant will be required to bring their current oral care products to Visit 1 for staff to verify the absence of known anti-sensitivity ingredients and DH claims.
* Participant who has had a professional de-sensitizing treatment within 8 weeks of Screening (Visit 1).
* Participant who habitually rinses with water during toothbrushing (self-reported at Screening Visit 1).
* Participant who seen to rinse with water while brushing with the acclimatization toothpaste during review of their brushing compliance videos at Baseline (Visit 2).
* Participant with known or suspected intolerance or hypersensitivity to the study products or any of their stated ingredients (or closely related compounds).
* Participant who is unwilling or unable to comply with product usage instructions or Lifestyle Considerations as described in the protocol.
* Female participant who is pregnant or intending to become pregnant during the study (self-reported).
* Female participant who is breastfeeding.
* Participant with a recent history (within the last year) of alcohol and/or substance abuse.
* Participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* Participant taking daily doses of medications or traditional herbal treatments which, in the opinion of the investigator or medically qualified designee, could interfere with their perception of pain.

  1. Examples of such medications include analgesics, anticonvulsants, antihistamines that cause marked or moderate sedation, sedatives, tranquilisers, anti-depressants, mood altering and anti-inflammatory drugs.
  2. Examples of herbal treatments include clove oil, olive oil or other treatments directly applied to the oral cavity for the treatment of oral health conditions.
* Participant taking daily doses of a medication which, in the opinion of the investigator or medically qualified designee, is causing xerostomia.
* Participant who requires antibiotic prophylaxis for dental procedures.
* At Screening (Visit 1): participant who has taken antibiotics within 2 weeks of their Screening visit.
* At Baseline (Visit 2): participant who has taken antibiotics within 2 weeks of their Baseline visit (during the acclimatisation period).
* Participant who has had a professional or self-applied tooth bleaching procedure within 8 weeks of Screening (Visit 1).
* Participant who has had dental prophylaxis within 4 weeks of Screening (Visit 1).
* Participant who has had treatment for periodontal disease (including surgery) within 12 months of Screening (Visit 1).
* Participant who has had scaling or root planning within 3 months of Screening (Visit 1).
* Participant with a tongue or lip piercing.
* Participant with, in the opinion of the investigator or medically qualified designee, gross periodontal disease.
* Participant with evidence of gross intra-oral neglect or the need for extensive dental therapy.
* Participant with a fixed or removable partial prosthesis which, in the opinion of the investigator or medically qualified designee, would impact study outcomes.
* Participant with multiple dental implants which, in the opinion of the investigator or medically qualified designee, would impact study outcomes.
* Participant with fixed or removable orthodontic braces/bands or a fixed orthodontic retainer.
* Participant with specific dentition exclusions for "Test Teeth" are as follows:

  1. Tooth with evidence of current or recent caries or reported treatment of decay within 12 months of Screening (Visit 1).
  2. Tooth with exposed dentin but with deep, defective or facial restorations.
  3. Tooth with full crown or veneer.
  4. Tooth adjacent to a bridge abutment or crown which, in the opinion of the investigator or medically qualified designee, would impact study outcomes.
  5. Sensitive tooth with contributing aetiologies other than erosion, abrasion or recession to exposed dentine.
  6. Sensitive tooth, in the opinion of the investigator or medically qualified designee, not expected to respond to treatment with an anti-sensitivity toothpaste.
* Participant who has previously been enrolled in this study.
* Any participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2023-09-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Preventive Dentistry, Shanghai Ninth People's Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center in China.
Pre-assignment Details: A total of 720 participants were screened of which 416 participants were enrolled and 243 participants were randomized to receive treatment in 3 groups - Test group (97 participants), Positive Control group (50 participants) and Negative Control group (96 participants). A total of 240 randomized participants completed the study.
Groups:
- Test Dentifrice (Sensodyne Sensitivity and Gum): Participants brushed the two test teeth first, then the whole mouth (all teeth) with Sensodyne Sensitivity and Gum toothpaste containing 0.454 percent (%) weight by weight (w/w) Stannous fluoride (SnF2) for 1-timed minute, twice daily (morning and evening) for up to 12 weeks. After brushing, participants rinsed once with 10 milliliters (mL) of water using the measuring cup provided.
- Positive Control (Sensodyne Repair and Protect): Participants brushed the two test teeth first, then the whole mouth (all teeth) with Sensodyne Repair and Protect toothpaste containing 5.0% w/w Calcium sodium phosphosilicate (CSPS) for 1-timed minute, twice daily (morning and evening) for up to 12 weeks. After brushing, participants rinsed once with 10 mL of water using the measuring cup provided.
- Negative Control (Crest Cavity Protection Fresh Lime): Participants brushed the two test teeth first, then the whole mouth (all teeth) with Crest Cavity Protection Fresh Lime toothpaste (regular fluoride toothpaste) for 1-timed minute, twice daily (morning and evening) for up to 12 weeks. After brushing, participants rinsed once with 10 mL of water using the measuring cup provided.
Period: Overall Study
Arm/Group | Test Dentifrice (Sensodyne Sensitivity and Gum) | Positive Control (Sensodyne Repair and Protect) | Negative Control (Crest Cavity Protection Fresh Lime)
Started | 97 | 50 | 96
Completed | 95 | 49 | 96
Not Completed | 2 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Modified Intent-To-Treat (mITT) population included all randomized participants who completed at least one use of study product and had at least one post-Baseline efficacy assessment.
Groups:
- Test Dentifrice (Sensodyne Sensitivity and Gum): Participants brushed the two test teeth first, then the whole mouth (all teeth) with Sensodyne Sensitivity and Gum toothpaste containing 0.454% w/w SnF2 for 1-timed minute, twice daily (morning and evening) for up to 12 weeks. After brushing, participants rinsed once with 10mL of water using the measuring cup provided.
- Positive Control (Sensodyne Repair and Protect): Participants brushed the two test teeth first, then the whole mouth (all teeth) with Sensodyne Repair and Protect toothpaste containing 5.0% w/w CSPS for 1-timed minute, twice daily (morning and evening) for up to 12 weeks. After brushing, participants rinsed once with 10 mL of water using the measuring cup provided.
- Total: Total of all reporting groups
Arm/Group | Test Dentifrice (Sensodyne Sensitivity and Gum) | Positive Control (Sensodyne Repair and Protect) | Negative Control (Crest Cavity Protection Fresh Lime) | Total
Number analyzed (Participants) | 95 | 49 | 96 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (7.64) | 43.7 (7.55) | 43.2 (7.57) | 43.0 (7.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 47 | 88 | 224
  Male | 6 | 2 | 8 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - East Asian Heritage | 95 | 49 | 96 | 240

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in Schiff Sensitivity Score (Average of the Two Selected Test Teeth) at Week 12 (Test Dentifrice Versus [vs.] Negative Control)
Description: Schiff sensitivity score was assessed by participant's response to an evaporative (air) stimulus after the stimulation of the 2 test teeth selected at Baseline by the examiner. Participant's response was scored using Schiff sensitivity scale, an examiner-based index, scored immediately following administration of the evaporative (air) stimulus. Score ranged from 0-3 where 0=Participant did not respond to air stimulation; 1=Participant responded to air stimulus but did not request discontinuation of stimulus; 2=Participant responded to air stimulus and requested discontinuation or moved from stimulus; 3=Participant responded to stimulus, considered stimulus to be painful, and requested discontinuation of the stimulus. Higher score indicated worse outcome (more sensitivity). Change from Baseline was calculated by subtracting the Baseline value from the value at indicated timepoint. Baseline was defined as Day 1 value. A negative change from Baseline indicated improvement in sensitivity.
Time Frame: Baseline and Week 12
Population: mITT population.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Test Dentifrice (Sensodyne Sensitivity and Gum): Participants brushed the two test teeth first, then the whole mouth (all teeth) with Sensodyne Sensitivity and Gum toothpaste containing 0.454% w/w SnF2 for 1-timed minute, twice daily (morning and evening) for up to 12 weeks. After brushing, participants rinsed once with 10 mL of water using the measuring cup provided.
Arm/Group | Test Dentifrice (Sensodyne Sensitivity and Gum) | Negative Control (Crest Cavity Protection Fresh Lime)
Number analyzed (Participants) | 95 | 96
score on a scale | -0.90 (0.068) | -0.74 (0.068)
Statistical Analysis 1: Comparison: Test Dentifrice (Sensodyne Sensitivity and Gum) vs Negative Control (Crest Cavity Protection Fresh Lime); Test type: Superiority; p = 0.0871, Mixed Model with Repeated Measure (MMRM); Adjusted Mean Difference = -0.17, 95% CI 2-sided [-0.36 to 0.02], Standard Error of Mean 0.096 — Adjusted mean difference was calculated as test minus negative control

2. Secondary Outcome: Adjusted Mean Change From Baseline in Tactile Threshold (Gram [g]) (Average of the Two Selected Test Teeth) at Week 12 (Test Dentifrice vs. Negative Control)
Description: Tactile sensitivity was assessed for eligible incisor, canine and pre-molar teeth using a constant pressure probe (Yeaple probe). The probe tip was placed perpendicular to the facial surface of tooth and drawn slowly across the exposed dentine. After each application of the stimulus, the participant was asked to indicate whether they experienced any pain or discomfort (yes/no response). The pressure setting with two consecutive 'yes' responses was recorded as the tactile threshold (g). At Baseline, the upper force setting was 20 g. Tactile threshold (g) was derived as the mean value for the two 'Test Teeth' selected by the examiner at Baseline. Higher tactile threshold indicated better outcome (less sensitivity). Change from Baseline was calculated by subtracting Baseline value from the value at indicated timepoint. Baseline was defined as Day 1 value. A positive change from Baseline indicated an improvement in sensitivity.
Time Frame: Baseline and Week 12
Population: mITT population.
Measure: Mean (Standard Error); unit: grams
Arm/Group | Test Dentifrice (Sensodyne Sensitivity and Gum) | Negative Control (Crest Cavity Protection Fresh Lime)
Number analyzed (Participants) | 95 | 96
grams | 25.86 (3.008) | 19.65 (2.977)
Statistical Analysis 1: Comparison: Test Dentifrice (Sensodyne Sensitivity and Gum) vs Negative Control (Crest Cavity Protection Fresh Lime); Test type: Superiority; p = 0.0972, van Elteren Test; P-value was from the van Elteren test adjusted for Baseline Schiff sensitivity stratification factor; Adjusted Mean Difference = 6.21, 95% CI 2-sided [-0.78 to 13.20], Standard Error of Mean 3.548 — Adjusted mean difference was calculated as test minus negative control

3. Secondary Outcome: Adjusted Mean Change From Baseline in Visual Analog Scale (VAS) Score (Millimeters [mm]) (Average of the Two Selected Test Teeth) at Week 12 (Test Dentifrice vs. Negative Control)
Description: Evaporative (air) sensitivity was assessed on the facial surfaces of the two test teeth selected by the examiner at Baseline by directing a 1 second application of air from standard dental syringe held perpendicular to tooth surface. Participant's response to the stimulus was evaluated using Schiff sensitivity scale with scores ranging from 0 (Participant did not respond to air stimulation) to 3 (Responded to stimulus, considered stimulus to be painful, requested discontinuation of the stimulus). Participants then rated the intensity of their response to the evaporative (air) stimulus using a 100 mm VAS with scores ranging from 0 mm (No discomfort) to 100 mm (Extreme discomfort; worst imaginable). Higher score indicated worse outcome (higher sensitivity). Change from Baseline was calculated by subtracting Baseline value from the value at indicated timepoint. Baseline was defined as Day 1 value. A negative change from Baseline indicated an improvement in sensitivity.
Time Frame: Baseline and Week 12
Population: mITT population.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Test Dentifrice (Sensodyne Sensitivity and Gum) | Negative Control (Crest Cavity Protection Fresh Lime)
Number analyzed (Participants) | 95 | 96
score on a scale | -38.84 (2.872) | -33.02 (2.830)
Statistical Analysis 1: Comparison: Test Dentifrice (Sensodyne Sensitivity and Gum) vs Negative Control (Crest Cavity Protection Fresh Lime); Test type: Superiority; p = 0.0671, MMRM; Adjusted Mean Difference = -5.81, 95% CI 2-sided [-12.04 to 0.41], Standard Error of Mean 3.160 — Adjusted mean difference was calculated as test minus negative control

4. Secondary Outcome: Adjusted Mean Change From Baseline in Schiff Sensitivity Score (Average of the Two Selected Test Teeth) at Week 6 (Test Dentifrice vs. Negative Control)
Description: as for outcome 1
Time Frame: Baseline and Week 6
Population: mITT population. Only those participants with data available at the indicated timepoint were analyzed.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Test Dentifrice (Sensodyne Sensitivity and Gum) | Negative Control (Crest Cavity Protection Fresh Lime)
Number analyzed (Participants) | 93 | 95
score on a scale | -0.51 (0.049) | -0.38 (0.049)
Statistical Analysis 1: Comparison: Test Dentifrice (Sensodyne Sensitivity and Gum) vs Negative Control (Crest Cavity Protection Fresh Lime); Test type: Superiority; p = 0.0673, MMRM; Adjusted Mean Difference = -0.13, 95% CI 2-sided [-0.27 to 0.01], Standard Error of Mean 0.070 — Adjusted mean difference was calculated as test minus negative control

5. Secondary Outcome: Adjusted Mean Change From Baseline in Tactile Threshold (g) (Average of the Two Selected Test Teeth) at Week 6 (Test Dentifrice vs. Negative Control)
Description: Tactile sensitivity was assessed for eligible incisor, canine and pre-molar teeth using a constant pressure probe (Yeaple probe). The probe tip was placed perpendicular to the facial surface of tooth and drawn slowly across the exposed dentine. After each application, the participant was asked to indicate whether they experienced any pain or discomfort (yes/no response). The pressure setting with two consecutive 'yes' responses was recorded as the tactile threshold (g). At Baseline, the upper force setting was 20 g. Tactile threshold (g) was derived as the mean value for the two 'Test Teeth' selected by the examiner at Baseline. Higher tactile threshold indicated better outcome (less sensitivity). Change from Baseline was calculated by subtracting Baseline value from the value at indicated timepoint. Baseline was defined as Day 1 value. A positive change from Baseline indicated an improvement in sensitivity.
Time Frame: Baseline and Week 6
Population: mITT population. Only those participants with data available at the indicated timepoint were analyzed.
Measure: Mean (Standard Error); unit: grams
Arm/Group | Test Dentifrice (Sensodyne Sensitivity and Gum) | Negative Control (Crest Cavity Protection Fresh Lime)
Number analyzed (Participants) | 93 | 95
grams | 11.74 (2.393) | 9.36 (2.357)
Statistical Analysis 1: Comparison: Test Dentifrice (Sensodyne Sensitivity and Gum) vs Negative Control (Crest Cavity Protection Fresh Lime); Test type: Superiority; p = 0.4050, van Elteren Test; P-value was from the van Elteren test adjusted for Baseline Schiff sensitivity stratification factor; Adjusted Mean Difference = 2.38, 95% CI 2-sided [-2.44 to 7.20], Standard Error of Mean 2.446 — Adjusted mean difference was calculated as test minus negative control

6. Secondary Outcome: Adjusted Mean Change From Baseline in VAS Score (mm) (Average of the Two Selected Test Teeth) at Week 6 (Test Dentifrice vs. Negative Control)
Description: Evaporative (air) sensitivity was assessed on the facial surfaces of the two test teeth selected by the examiner at Baseline by directing a 1 second application of air from standard dental syringe held perpendicular to tooth surface. Participant's response to the stimulus was evaluated using Schiff sensitivity scale with scores ranging from 0 (Participant did not respond to air stimulation) to 3 (Responded to stimulus, considered stimulus to be painful, requested discontinuation of the stimulus). Participant then rated the intensity of their response to the evaporative (air) stimulus using a 100 mm VAS with scores ranging from 0 mm (No discomfort) to 100 mm (Extreme discomfort; worst imaginable). Higher score indicated worse outcome (higher sensitivity). Change from Baseline was calculated by subtracting Baseline value from the value at indicated timepoint. Baseline was defined as Day 1 value. A negative change from Baseline indicated an improvement in sensitivity.
Time Frame: Baseline and Week 6
Population: mITT population. Only those participants with data available at the indicated timepoint were analyzed.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Test Dentifrice (Sensodyne Sensitivity and Gum) | Negative Control (Crest Cavity Protection Fresh Lime)
Number analyzed (Participants) | 93 | 95
score on a scale | -21.92 (2.603) | -16.28 (2.556)
Statistical Analysis 1: Comparison: Test Dentifrice (Sensodyne Sensitivity and Gum) vs Negative Control (Crest Cavity Protection Fresh Lime); Test type: Superiority; p = 0.0346, MMRM; Adjusted Mean Difference = -5.64, 95% CI 2-sided [-10.88 to -0.41], Standard Error of Mean 2.656 — Adjusted mean difference was calculated as test minus negative control

7. Secondary Outcome: Adjusted Mean Change From Baseline in Schiff Sensitivity Score (Average of the Two Selected Test Teeth) at Week 6 and Week 12 (Positive Control vs. Negative Control)
Description: as for outcome 1
Time Frame: Baseline, Week 6 and Week 12
Population: mITT population. Only those participants with data available at the indicated timepoints were analyzed.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Positive Control (Sensodyne Repair and Protect) | Negative Control (Crest Cavity Protection Fresh Lime)
Number analyzed (Participants) | 49 | 96
score on a scale
  Change from Baseline at Week 6: number analyzed (Participants) | 47 | 95
  Change from Baseline at Week 6 | -0.36 (0.069) | -0.38 (0.049)
  Change from Baseline at Week 12 | -0.67 (0.095) | -0.74 (0.068)
Statistical Analysis 1: Comparison: Positive Control (Sensodyne Repair and Protect) vs Negative Control (Crest Cavity Protection Fresh Lime); Change from Baseline at Week 6; Test type: Superiority; p = 0.8256, MMRM; Adjusted Mean Difference = 0.02, 95% CI 2-sided [-0.15 to 0.19], Standard Error of Mean 0.085 — Adjusted mean difference was calculated as positive control minus negative control
Statistical Analysis 2: Comparison: Positive Control (Sensodyne Repair and Protect) vs Negative Control (Crest Cavity Protection Fresh Lime); Change from Baseline at Week 12; Test type: Superiority; p = 0.5314, MMRM; Adjusted Mean Difference = 0.07, 95% CI 2-sided [-0.16 to 0.30], Standard Error of Mean 0.117 — Adjusted mean difference was calculated as positive control minus negative control

8. Secondary Outcome: Adjusted Mean Change From Baseline in Tactile Threshold (g) (Average of the Two Selected Test Teeth) at Week 6 and Week 12 (Positive Control vs. Negative Control)
Description: Tactile sensitivity was assessed for eligible incisor, canine and pre-molar teeth using a constant pressure probe (Yeaple probe). The probe tip was placed perpendicular to the facial surface of tooth and drawn slowly across the exposed dentine. After each application of the stimulus, the participant was asked to indicate whether they experienced any pain or discomfort (yes/no response). The pressure setting with two consecutive 'yes' responses was recorded as the tactile threshold (g). At Baseline, the upper force setting was 20 g. Tactile threshold (g) was derived as the mean value for the two 'Test Teeth' selected by the examiner at Baseline. Higher tactile threshold indicated better outcome (less sensitivity). Change from Baseline was calculated by subtracting Baseline value from the value at indicated timepoint. Baseline was defined as Day 1 value. A positive change from Baseline indicated an improvement.
Time Frame: Baseline, Week 6 and Week 12
Population: mITT population. Only those participants with data available at the indicated timepoints were analyzed.
Measure: Mean (Standard Error); unit: grams
Arm/Group | Positive Control (Sensodyne Repair and Protect) | Negative Control (Crest Cavity Protection Fresh Lime)
Number analyzed (Participants) | 49 | 96
grams
  Change from Baseline at Week 6: number analyzed (Participants) | 47 | 95
  Change from Baseline at Week 6 | 6.77 (2.883) | 9.36 (2.357)
  Change from Baseline at Week 12 | 18.53 (3.830) | 19.65 (2.977)
Statistical Analysis 1: Comparison: Positive Control (Sensodyne Repair and Protect) vs Negative Control (Crest Cavity Protection Fresh Lime); Change from Baseline at Week 6; Test type: Superiority; p = 0.5575, van Elteren Test; P-value was from the Van Elteren test adjusted for Baseline Schiff sensitivity stratification factor; Adjusted Mean Difference = -2.59, 95% CI 2-sided [-8.48 to 3.30], Standard Error of Mean 2.990 — Adjusted mean difference was calculated as positive control minus negative control
Statistical Analysis 2: Comparison: Positive Control (Sensodyne Repair and Protect) vs Negative Control (Crest Cavity Protection Fresh Lime); Change from Baseline at Week 12; Test type: Superiority; p = 0.7717, van Elteren Test; P-value was from the van Elteren test adjusted for Baseline Schiff sensitivity stratification factor; Adjusted Mean Difference = -1.12, 95% CI 2-sided [-9.60 to 7.37], Standard Error of Mean 4.308 — Adjusted mean difference was calculated as positive control minus negative control

9. Secondary Outcome: Adjusted Mean Change From Baseline in VAS Score (mm) (Average of the Two Selected Test Teeth) at Week 6 and Week 12 (Positive Control vs. Negative Control)
Description: Evaporative (air) sensitivity was assessed on the facial surfaces of the two test teeth selected by the examiner at Baseline by directing a 1 second application of air from standard dental syringe held perpendicular to tooth surface. Participant's response to the stimulus was evaluated using Schiff sensitivity scale with scores ranging from 0(Participant did not respond to air stimulation) to 3(Responded to stimulus, considered stimulus to be painful, requested discontinuation of the stimulus). Participant then rated the intensity of their response to the evaporative (air) stimulus using a 100 mm VAS with scores ranging from 0 mm (No discomfort) to 100 mm (Extreme discomfort; worst imaginable). Higher score indicated worse outcome (higher sensitivity). Change from Baseline was calculated by subtracting Baseline value from the value at indicated timepoint. Baseline was defined as Day 1 value. A negative change from Baseline indicated an improvement in sensitivity.
Time Frame: Baseline, Week 6 and Week 12
Population: mITT population. Only those participants with data available at the indicated timepoints were analyzed.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Positive Control (Sensodyne Repair and Protect) | Negative Control (Crest Cavity Protection Fresh Lime)
Number analyzed (Participants) | 49 | 96
score on a scale
  Change from Baseline at Week 6: number analyzed (Participants) | 47 | 95
  Change from Baseline at Week 6 | -15.53 (3.123) | -16.28 (2.556)
  Change from Baseline at Week 12 | -29.30 (3.542) | -33.02 (2.830)
Statistical Analysis 1: Comparison: Positive Control (Sensodyne Repair and Protect) vs Negative Control (Crest Cavity Protection Fresh Lime); Change from Baseline at Week 6; Test type: Superiority; p = 0.8180, MMRM; Adjusted Mean Difference = 0.75, 95% CI 2-sided [-5.63 to 7.12], Standard Error of Mean 3.235 — Adjusted mean difference was calculated as positive control minus negative control
Statistical Analysis 2: Comparison: Positive Control (Sensodyne Repair and Protect) vs Negative Control (Crest Cavity Protection Fresh Lime); Change from Baseline at Week 12; Test type: Superiority; p = 0.3322, MMRM; Adjusted Mean Difference = 3.73, 95% CI 2-sided [-3.83 to 11.28], Standard Error of Mean 3.834 — Adjusted mean difference was calculated as positive control minus negative control

ADVERSE EVENTS:
Time Frame: From signing of the informed consent form until 5 days following the last administration of the study product or last study procedure (up to approximately 123 days).
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study product including any washout or lead-in product (or medical device), whether or not considered related to the study product, including any washout or lead-in product. All-Cause Mortality included all randomized participants. Serious and Other AEs: Safety population included all participants who completed at least one use of study product.
Arm/Group | Test Dentifrice (Sensodyne Sensitivity and Gum) | Positive Control (Sensodyne Repair and Protect) | Negative Control (Crest Cavity Protection Fresh Lime)
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/50 | 0/96
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/50 | 0/96
Other Adverse Events (participants affected / at risk) | 16/97 | 9/50 | 11/96
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Dentifrice (Sensodyne Sensitivity and Gum) (N=97) | Positive Control (Sensodyne Repair and Protect) (N=50) | Negative Control (Crest Cavity Protection Fresh Lime) (N=96)
LIP ULCERATION (Gastrointestinal disorders) | 1 | 0 | 2
MOUTH ULCERATION (Gastrointestinal disorders) | 3 | 0 | 0
ANGULAR CHEILITIS (Gastrointestinal disorders) | 2 | 0 | 0
ORAL BLOOD BLISTER (Gastrointestinal disorders) | 0 | 0 | 2
CHEILITIS (Gastrointestinal disorders) | 1 | 0 | 0
DENTAL CARIES (Gastrointestinal disorders) | 0 | 0 | 1
ORAL CAVITY FISTULA (Gastrointestinal disorders) | 0 | 1 | 0
ORAL MUCOSAL BLISTERING (Gastrointestinal disorders) | 0 | 1 | 0
TONGUE ULCERATION (Gastrointestinal disorders) | 1 | 0 | 0
MOUTH INJURY (Injury, poisoning and procedural complications) | 3 | 2 | 1
FACE INJURY (Injury, poisoning and procedural complications) | 0 | 2 | 1
LIP INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0
PALATE INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
GINGIVITIS (Infections and infestations) | 2 | 1 | 0
GINGIVAL ABSCESS (Infections and infestations) | 0 | 1 | 1
ABSCESS ORAL (Infections and infestations) | 0 | 0 | 1
HERPES SIMPLEX (Infections and infestations) | 0 | 1 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 0 | 1
PERIODONTITIS (Infections and infestations) | 1 | 0 | 0
MUCOSAL INFLAMMATION (General disorders) | 1 | 0 | 0
OEDEMA MUCOSAL (General disorders) | 0 | 1 | 0
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
BLOOD BLISTER (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
HALEON agreements may vary with individual investigators but will not prohibit any investigator from publishing. HALEON supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/45/NCT05750745/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT05750745/SAP_001.pdf